CLINICAL TRIAL: NCT01994655
Title: Chinese Health Ivvestigation Of Nurse Aging
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bai Wen-Pei (Other)
Responsible Party: Sponsor-Investigator, Bai Wen-Pei, Peking University, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: PEK-8357-wp
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Hot Flashes
Keywords: climacteric symptoms; menopause; nurses
MeSH Terms: conditions — Hot Flashes | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doing exercise (Experimental): We want to use Kupperman Index to assess the severity of climacteric symptoms,and assess the effect of doing exercise fof the climacteric symptoms
  Interventions: Other: Doing exercise

INTERVENTIONS:
Other: Doing exercise — We want to investigate the effects of exercise on climacteric symptoms
  Other Names: Exercise
Other: Doing exercise — Doing exercise at least 6 months including walking, running, yoga etc.
  Other Names: Exercise

SUMMARY:
Climacteric symptoms can be treated by doing exercise,not hormone replacement therapy.

DETAILED DESCRIPTION:
Hormone replacement therapy(HRT) is the main therapy to climacteric symptoms. But HRT also has a lot of disadvantages, such as cardiovascular disease, breast cancer .In our previous investigation,we found that doing exercise is helpful for climacteric symptoms.So we want to make a detailed investigation to research it.

ELIGIBILITY:
Inclusion Criteria:

- Women aged 40-55 who has climacteric symptoms

Exclusion Criteria:

- Women who have serious climacteric symptoms and other diseases which could interrupt the research.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2008-08; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
KMI | up to 2 years
  KMI is the short of Kupperman Index,which is a questionnaire to assesses the severity of climacteric symptoms.

SECONDARY OUTCOMES:
blood lipid | up to 2 years
  Blood lipid is an index to assess the effect of doing exercise.